CLINICAL TRIAL: NCT06999616
Title: Promoting Physical Activity in Individuals With Cancer in an Oncology Day Clinic - Testing the Feasibility of the Implementation of a Physical Activity Concept Within an Interprofessional Team Led by Nurses OnkoMoveNurse - Proof of Concept
Brief Title: Physical Activity in Cancer Patients in an Oncology Day Clinic - Implementing a Person-centered Program Led by Nurses
Acronym: OnkoMoveNurse
Status: Recruiting | Type: Observational
Sponsor: St.Gallen University of Applied Sciences (Other)
Collaborators: Kantonsspital Münsterlingen (Other)
Responsible Party: Sponsor
Other Study IDs: OnkoMoveNurse-proof of concept
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-05

CONDITIONS: Neoplasms; Motor Activity; Chemotherapy; Antitumor Drugs; Activity Level
Keywords: activity promotions; proof-of-concept; implementation; activity concept; excercise; cancer patient; physical activity
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with cancer in oncology day clinic: patients who receive activity promoting during care at oncology day clinic

SUMMARY:
Background: Physical activity has demonstrated benefits in alleviating side effects and improving well-being in people with cancer. However, activity levels remain low during systemic treatment. Nurses are optimally positioned to lead interventions fostering an activity-friendly culture.

Objective: This study aims to evaluate the feasibility and potential effects of the nurse-led, interprofessionally developed physical activity concept OncoMoveNurse in an outpatient oncology setting.

Methods: Using a mixed-methods design over 15 months (10/2024-12/2025), the study includes implementation and evaluation phases. Quantitative data (n=50 patients, collected from 06/2025-09/2025) will assess primary (physical activity behavior) and secondary outcomes (self-efficacy, well-being, mood) via validated PROMs. Qualitative insights will be gathered through digital storytelling (n=2 patients, n=2 nurses) and one focus group (n=8 interprofessional team members). Inclusion criteria for patients include age ≥18, cancer diagnosis, at least three treatments in the day clinic, and sufficient German language skills.

Intervention: OncoMoveNurse comprises five adaptable components: modular activity structure, safety framework, communication strategy, a team approach, and person-centered orientation. Supporting materials (e.g., posters, videos, exercise tools) and tailored implementation strategies were co-developed in alignment with core values.

Analysis: Quantitative data will be analyzed using SPSS (paired t-tests, p<.05); qualitative data via content analysis in MAXQDA. A mixed-methods synthesis will integrate findings.

Ethics & Data Protection: Patient data collection will commence following ethics approval. All data are anonymized, stored securely, and handled in accordance with Swiss data protection laws.

Conclusion: This study will provide insights into the feasibility of nurse-led physical activity promotion in outpatient oncology and inform future outcome evaluations.

DETAILED DESCRIPTION:
Background and Rationale Staying physically active during cancer treatment can help alleviate distressing symptoms such as fatigue, pain, and dyspnoea, and can improve the quality of life of individuals with cancer. Nevertheless, physical activity often decreases during treatment due to various factors, including general physical decline, treatment-related side effects (e.g., nausea, dizziness, muscle weakness), and psychological factors (e.g., anxiety, lack of motivation, depressive symptoms). Other contributing factors may include breathlessness, oxygen deficiency, and reduced physical endurance.

To counteract this, individuals with cancer should be specifically encouraged to engage in physical activity during their outpatient visits-before, during, and after chemotherapy, immunotherapy, or other treatments. The goal is to integrate more physical activity into everyday life.

For this purpose, a dedicated physical activity concept has been developed by a team of experienced professionals. This concept is built around five core components:

1. A modular exercise catalogue
2. A safety protocol
3. A communication strategy
4. Team orientation
5. Person-centeredness Further details are available at www.onkomovenurse.net.

   ________________________________________ Risk / Benefit Assessment

   Benefits:

   Participants will not experience direct benefits from the survey. However, their involvement contributes to the improvement of clinical practice and scientific knowledge.

   At the personal level:

   Participants may experience improved well-being and reduced symptom burden (e.g., fatigue, pain, dyspnea). They will also receive support from oncology nurses to expand their repertoire of safe, low-threshold physical activity options.

   At the organizational level:

   Development of a practice-oriented physical activity concept tailored to patients and professionals; promotion of interprofessional collaboration; strengthening of the nursing role; enhancement of person-centered care and institutional reputation.

   At the research level:

   Systematic evaluation of the physical activity concept to improve care for individuals with cancer; strengthening the role of nurses in health promotion in the outpatient setting.

   Vision:

   To serve as a national model for symptom management and physical activity interventions in oncology care across Switzerland.

   ________________________________________ Objective(s) The aim of the project is to implement the OnkoMoveNurse physical activity concept in an oncology outpatient setting under the leadership of oncology nurses and to assess its feasibility for individuals with cancer. Quantitative and qualitative surveys of patients and healthcare professionals will provide initial insights into the potential effects on physical activity behaviour.

   ________________________________________ Endpoint(s) Primary endpoint: Physical activity behaviour of participants Secondary endpoints: Self-efficacy regarding physical activity, well-being, and mood. Demographic and clinical data will be collected to describe the sample.

   ________________________________________ Study Design Mixed-methods design

   ________________________________________ Inclusion / Exclusion Criteria Patients
   1. For the quantitative survey, n=50 patients will be invited who meet the following criteria:

      (1) diagnosis of cancer, (2) at least three treatments at the oncology outpatient clinic in Münsterlingen during the study period, (3) aged ≥18 years, and (4) sufficient knowledge of German. Pregnant individuals are excluded.
   2. For digital storytelling, n=2 patients will be recruited who meet the following criteria:

      (1) diagnosis of cancer, (2) currently undergoing systemic therapy in the collaborating oncology outpatient clinic, (3) aged ≥18 years, (4) sufficient knowledge of German, (5) willingness to use a mobile device (e.g., smartphone, tablet) for digital storytelling, and (6) not a member of the internal quality circle. Healthcare Professionals and Organization

   <!-- -->

   1. For digital storytelling, the following professionals will be recruited:

   i. n=2 oncology nurses employed in the outpatient clinic who care for individuals with cancer. One may be a project team member, while the other may not be directly involved in implementation.

   b. For a focus group interview, the following will be recruited: i. n=3 oncology nurses working in the oncology outpatient clinic, ii. n=2 physicians involved in cancer care in the same setting, iii. n=3 additional healthcare professionals (e.g., nursing assistants, reception staff, internal transport services).

   ________________________________________ Number of Participants with Rationale

   Quantitative survey:

   n=50 patients with cancer

   Digital storytelling:

   Total n=4
   * n=2 oncology nurses
   * n=2 patients with cancer

   Focus group interview:

   Total n=8

   - n=3 oncology nurses
   * n=2 physicians
   * n=3 other healthcare professionals (e.g., assistants, psycho-oncologists, reception or transport staff)

   Study Intervention The implementation of the OnkoMoveNurse physical activity concept in an oncology outpatient clinic will be evaluated using a mixed-methods study design. The study will span 15 months (10/2024-12/2025) and consist of three phases: preparation, implementation, and evaluation.

   The preparation phase has already started. A project group was established with support from the OST staff. Necessary materials have been developed and installed in the outpatient clinic to be used by all patients who pass a safety screening.

   Implementation will be led by the project group, OST collaborators, and clinic staff. Training sessions and seminars are planned, alongside opportunities for experiential learning and feedback. Upon completion, the project group will transition into a permanent "Physical Activity Quality Circle." Evaluation will begin after ethical approval and will involve collecting both quantitative and qualitative data from patients and healthcare professionals. Quantitative data will be collected via Patient-Reported Outcome Measures (PROMs). Qualitative data will be obtained through digital storytelling (a method previously used successfully in a large study), as well as personal interviews and feedback questionnaires.

   ________________________________________ Control Intervention N/A

   ________________________________________ Study Procedures The entire study period covers 15 months. Project start and preparation began on 01/10/2024. Implementation commenced on 19/02/2025. Evaluation research will begin upon receipt of ethical approval.

   ________________________________________ Study Duration and Schedule

   Estimated duration from first participant screened to last participant last visit:
   * First Participant In: Health care professionals 03/2025 / patients planned for 06/2025
   * Last Participant Out: Planned for 12/2025 / patients planned for 09/2025 Statistical Considerations Quantitative data will be analyzed using SPSS (version 28.0) following an intention-to-treat approach. Paired t-tests will be used (significance level: 0.05). Quality control measures include double-checking, data cleaning, and outlier analysis.

   Qualitative data from interviews and digital storytelling will be anonymized, transcribed, and analyzed using content analysis according to Kuckartz & Rädiker with MAXQDA 2024.

   The mixed-methods synthesis will integrate quantitative and qualitative results through thematic and statistical summaries to generate comprehensive findings.

   ________________________________________ Data Privacy All data will be stored and managed securely in accordance with data protection regulations.

   The research team affirms and ensures participants' rights to privacy and data protection, particularly in relation to the presentation of study results at scientific conferences or publication in journals.

   All relevant laws and guidelines, including the Swiss Federal Act on Data Protection (FADP), will be strictly followed.

   Individual medical information collected during the study will be treated as confidential and will not be disclosed to third parties. Access to study data will be restricted to authorized personnel involved in the project. Participant confidentiality will be ensured through assignment of a unique participant identification number (Patient ID).

   ________________________________________ Ethical Considerations All participants will receive comprehensive written and verbal information about the study, enabling them to provide informed consent before participating.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of cancer,
2. at least three treatments at the oncology outpatient clinic in Münsterlingen during the study period,
3. aged ≥18 years, and
4. sufficient knowledge of German.

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cancer patients who are treated at oncology day clinic
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
physical activity behaviour | from enrollment to the end of treatment or three months after enrollment whichever timepoint comes first
  Physical activity behavior will be assessed using the "Physical Activity and Sedentary Behavior Assessment Questionnaire" (BSA).
  The BSA consists of 16 items that capture the duration of physical activity in minutes per day across different intensity levels (light, moderate, vigorous), as well as daily sedentary time. Responses are aggregated and converted into minutes per week. The questionnaire demonstrates good internal consistency with Cronbach's alpha ranging from 0.82 to 0.89, and test-retest reliability of r = 0.76. Construct validity has been confirmed through correlations with accelerometer data (r = 0.68), and discriminant validity has been demonstrated by significant differences between active and inactive groups.

SECONDARY OUTCOMES:
Self-efficacy for physical activity | from enrollment to the end of treatment or three months after enrollment whichever timepoint comes first
  Self-efficacy for physical activity will be measured using the Self-Efficacy for Physical Activity Scale (SSA). The SSA assesses an individual's subjective belief in their ability to maintain regular physical activity despite potential barriers. The questionnaire comprises 12 items rated on a 7-point Likert scale, anchored by the verbal descriptors: not at all confident, maybe, and completely confident. The scale score for each participant is calculated as the arithmetic mean of all 12 item scores. The internal consistency of the SSA is high, with a Cronbach's alpha of 0.89 [36].
health-related quality of life | from enrollment to the end of treatment or three months after enrollment whichever timepoint comes first
  The EORTC QLQ-C30 is a standardized questionnaire used to assess health-related quality of life in individuals with cancer [37, 38].
  It consists of 30 items organized into five functional scales (physical, emotional, cognitive, social, and role functioning), three symptom scales (fatigue, pain, nausea/vomiting), a global health status/quality of life scale, and several single-item symptom measures. Responses are given on a four-point Likert scale (1 = not at all to 4 = very much). Scale scores are standardized, with higher scores on the functional scales indicating better quality of life.
  The internal consistency of the functional scales ranges from Cronbach's alpha = 0.70 to 0.90. The questionnaire demonstrates good test-retest reliability, as well as strong construct and criterion validity, and is widely used in oncological research.

CONTACTS AND LOCATIONS:
Overall Officials: Antje Koller, PhD, Principal Investigator — Eastern Switzerland University of Applied Sciences
Locations (1):
- Spital Thurgau AG Münsterlingen, Münsterlingen, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
fully anonymized data may be shared if interested researcher ensures proper handling of data
Supporting Information: Study Protocol
Time Frame: after study has been finished
Access Criteria: researchers may contact PI for more information